CLINICAL TRIAL: NCT02833207
Title: Peripheral Vasodilation in Obese Humans
Acronym: ObeseDilate
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to COVID-19, difficulty obtaining study drugs, difficulty recruiting obese subjects, and limited access to on-call physicians.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-0199; A176000 (Other: UW Madison); EDUC\KINESIOLOGY\KINESIO (Other: UW Madison); R01HL105820 (NIH); Protocol Version 4/27/2021 (Other: UW Madison)
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Obesity
Keywords: blood flow; vasodilation; Doppler Ultrasound; endothelium dependent dilation
MeSH Terms: conditions — Obesity; Aneurysm | interventions — UBR5 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- EDD Obese (Experimental): On study visit after screening. Brachial artery catheter in the non-dominant arm + infusion drugs (IND approval) to test basic vascular function and associated mechanisms in healthy volunteers. Eligible obese subjects will undergo Drug Trial 1 (EDD) (described in Intervention section).
  Interventions: Drug: Drug Trial 1 (EDD)
- EDD Lean (Experimental): On study visit after screening. Brachial artery catheter in the non-dominant arm + infusion drugs (IND approval) to test basic vascular function and associated mechanisms in healthy volunteers. Eligible lean subjects will undergo Drug Trial 1 (EDD) (described in Intervention section).
  Interventions: Drug: Drug Trial 1 (EDD)
- ROV Obese (Experimental): On study visit after screening. Brachial artery catheter in the non-dominant arm + infusion drugs (IND approval) to test basic vascular function and associated mechanisms in healthy volunteers. Eligible obese subjects will undergo Drug Trial 2 (ROV) (described in Intervention section).
  Interventions: Drug: Drug Trial 2 (ROV)
- ROV Lean (Experimental): On study visit after screening. Brachial artery catheter in the non-dominant arm + infusion drugs (IND approval) to test basic vascular function and associated mechanisms in healthy volunteers. Eligible lean subjects will undergo Drug Trial 2 (ROV) (described in Intervention section).
  Interventions: Drug: Drug Trial 2 (ROV)

INTERVENTIONS:
Drug: Drug Trial 1 (EDD) — Drugs that increase blood flow and test EDD are: ACh, ISO, BK, ATP. Remaining drugs used to test mechanisms of EDD: L-NMMA, ketorolac, and BaCl2.
  Details under study description.
  Other Names: EDD
  Arms: EDD Lean; EDD Obese
Drug: Drug Trial 2 (ROV) — Tools used to increase blood flow: muscle contractions and ATP. Remaining drugs used to test mechanisms of ROV: L-NMMA, ketorolac, and BaCl2.
  Details under study description.
  Other Names: ROV
  Arms: ROV Lean; ROV Obese

SUMMARY:
The growing population of obese adults is predicted to create a large public health burden in the next few decades. This study examines function of small blood vessels providing blood flow to skeletal muscles, to test if younger obese individuals (≤40 years old, BMI >30) are already displaying reductions in blood vessel function. This study will test if the signals blood vessels use to increase blood flow are changing in these same subjects. Findings from this study may help create treatments to delay or prevent some of the negative effects of obesity on vascular health.

DETAILED DESCRIPTION:
This study initially started in June 2011(IND 122211). The original Aim 1 was completed and showed lean and obese groups did not differ in endothelial dependent dilation (EDD) and exercise dilation responses. The original Aim 2 was contingent upon there being a difference between lean and obese groups in Aim 1 and therefore was not pursued.

The investigators now plan to continue this study by assessing 2 additional aims that are consistent with the original purpose of the study and are discussed below:

The growing population of obese adults is predicted to create a large public health burden in the next few decades. Obese humans also exhibit reduced exercise capacity and lower muscle blood flow. The overall goal of this research program is to investigate the obesity-related changes in microvascular function contributing to impaired muscle blood flow. This proposal seeks to directly test vascular control in human skeletal muscle resistance arteries in exercising humans. The investigators propose to study younger obese adults, without confounding effects of age, metabolic syndrome, or diabetes-before the negative effects of obesity can exert their full negative impact. The general hypothesis is that endothelium dependent dilation (EDD) and functional (exercise) vasodilation is impaired via shift away from nitric oxide bioavailability and a shift toward increased reliance on potassium (K+) mediated vasodilation.

Primary objective To determine whether role of K+ mediated vasodilation differs between lean and obese adults.

Aims Aim 1: To test the hypothesis that obesity induces an endothelial phenotype change that creates an environment for both EDD and exercise dysfunction. The investigators propose that obesity alters endothelial enzymes, which help explain the mechanistic changes in vasodilation.

Aim 2: To test the hypothesis that obesity elicits altered endothelial-dependent (EDD) and functional vasodilation due to altered functional potassium channel signaling. The investigators propose that potassium (K+) channel function accounts for unexplained differences in EDD and functional vasodilation. More specifically, the investigators hypothesize that inhibition of K+ mediated hyperpolarization (Inward Rectifying K+ channels-KIR) will identify differential vasodilator mechanisms between lean and obese adults.

Study Design and Overview of Procedures This study is designed to test cardiovascular control in clinically healthy humans. There will be 2 separate, scientifically distinct experimental trials that will be conducted in lean and obese subject: 1) EDD or 2) Rapid Onset Vasodilator (ROV), which studies the immediate increase in blood flow at the onset of exercise.

Common procedures between protocols: After screening to determine eligibility, subjects visit the lab for either EDD or Rapid Onset Vasodilator (ROV) study visit. All pre-screening and pre-visit procedures will be identical. A physician will place a brachial arterial catheter in the non-dominant arm for local drug infusion. Changes in blood flow will be quantified by Doppler ultrasound at the brachial artery. Monitoring of subject hemodynamics (Heart Rate, Blood Pressure, blood oxygen) is identical.

EDD experiments: EDD agonists are drugs than cause vasodilation to increase blood flow temporarily. The investigators will use 4 different agonists to test EDD function from several perspectives. After control EDD agonist infusions, subjects will repeat EDD agonists under conditions of K+ channel inhibition, and again under K+ channels plus nitric oxide and prostaglandin inhibition. This last phase of the study is aimed at testing acute compensatory/redundant vasodilator mechanisms. These trials will involve infusion of endothelial agonists, with and without inhibition of specific vasodilatory mechanisms. Agonists include: ATP, Bradykinin (BK), Isoproterenol (ISO), and Acetylcholine (Ach), will be infused 3 times each (order randomized). Agonists will be infused under the following conditions: 1) Alone (control) 2) in combination with Barium Chloride (BaCl2) 3) in combination with BaCl2, L-N-monomethyl Arginine Acetate (L-NMMA), and Ketorolac. EDD agonists each cause a temporary increase in forearm blood flow, which returns to baseline within minutes after infusion has stopped. Antagonists (BaCl2, L-NMMA and ketorolac) will likely reduce EDD responses to agonists, and may also reduce resting forearm blood flow or increase blood pressure (e.g. L-NMMA may decrease forearm blood flow 30-50% an increase BP 5-10 mmHg). The entire EDD study visit will be ~5 hours (1 hour setup and 4 hours experimental procedures). The EDD protocol is further described here:

Drugs (IND approval) are used to test basic science vascular function & associated mechanisms in healthy volunteers. Drugs not used to improve a health condition.

Drugs: acetylcholine, isoproterenol, bradykinin, adenosine triphosphate, barium chloride, L-N-monomethyl Arginine Acetate, ketorolac.

1. 5 minute saline infusion along with 2 minutes of ATP infusion,
2. 10 minute washout,
3. 5 minutes of saline solution along with 2 minutes of BK infusion,
4. 10 minute washout,
5. 5 minutes of saline solution along with 2 minutes of ISO infusion,
6. 10 minute washout,
7. 5 minutes of saline infusion along with 2 minutes of ACh infusion,
8. 10 minute washout,
9. 5 minutes of BaCl2 infusion and 2 minute of ATP infusion,
10. 10 minute washout,
11. 5 minutes of BaCl2 infusion along with 2 minutes of ACh infusion,
12. 10 minute washout,
13. 5 minutes of BaCl2 infusion along with 2 minutes of ISO infusion,
14. 10 minute washout,
15. 5 minutes of BaCl2 infusion along with 2 minutes of BK infusion,
16. 10 minute washout,
17. 10 minute L-NMMA and ketorolac infusion (continuous infusion throughout remainder of protocol) along with 5 minutes of BaCl2 infusion, and 2 minutes of ACh infusion,
18. 10 minute washout,
19. 5 minutes of BaCl2 infusion along with 2 minutes of ISO infusion,
20. 10 minute washout,
21. 5 minutes of BaCl2 infusion along with 2 minutes of ATP infusion,
22. 10 minute washout,
23. 5 minutes of BaCl2 infusion along with 2 minutes of BK infusion.

ROV experiments: After control single forearm muscle contractions, subjects will repeat single contractions under conditions of K+ channel inhibition, and again under K+ channel plus nitric oxide and prostaglandin inhibition. This last phase of the study is aimed at testing acute compensatory/redundant vasodilator mechanisms. This trial consists of three sets of 6 singular muscle contractions (three at 30%, three at 60% of maximal effort), each contraction lasting less than 3 seconds with ~90s rest in between. These single contractions evoke a robust (100-600% increase) and rapid (3-6 heart beats post contraction) increase in blood flow that returns to normal typically in about 30 seconds. This rapid and robust response is why these single muscle contractions are termed "Rapid Onset Vasodilation". 3 minutes of rest before each trial will allow for baseline measurements and loading of inhibitors of K+ mediated vasodilation. During this 3 min, subjects will perform a single contraction at 15, 30, and 45s of the 3-min loading/resting period to facilitate delivery of the drug to the active tissues (this adds an additional 18 contractions. The first experimental set of single contractions will be completed without drugs (saline control). Next, an ATP infusion (no exercise) will also be used to test the pharmacological efficacy of subsequent inhibitor (BaCl2). The first ATP infusion will be performed without other drugs. Following this, a second set of single contractions will be conducted with infusion of BaCl2. This is then followed by a second ATP infusion to determine the efficacy of BaCl2. The final set of single contractions will start and be performed with simultaneous infusion of all three inhibitors (BaCl2, L-NMMA, and Ketorolac). This last phase of the study is aimed at testing acute compensatory/redundant vasodilator mechanisms. ROV (exercise) studies will be ~4 hours (1 hour set up and 3 hours experimental procedures). The ROV protocol is further described here:

Drugs: adenosine triphosphate, barium chloride, L-N-monomethyl Arginine Acetate, ketorolac

1. 3 muscle contractions during 3 minute saline infusion followed by 3 additional muscle contractions,
2. Repeat 3 muscle contractions during 3 minute saline infusion followed by 3 additional muscle contractions ,
3. 10 minute washout,
4. Two minutes of ATP infusion,
5. 10 minute washout,
6. 3 muscle contractions during 3 minute BaCl2 infusion followed by 3 additional muscle contractions,
7. 3 muscle contractions during 3 minute BaCl2 infusion followed by 3 additional muscle contractions,
8. 10 minute washout,
9. Infusion of BaCl2 (3 minutes) and ATP (2 minutes),
10. 10 minute washout,
11. 3 muscle contractions during Infusion of BaCl2 (3 minutes) and L-NMMA and ketorolac infusion (5 minutes) followed by 3 additional muscle contractions,
12. L-NMMA and ketorolac will be infused throughout remainder of protocol at a lower dosage
13. 3 muscle contractions during Infusion of BaCl2 (3 minutes) and L-NMMA and ketorolac (5 minutes) followed by 3 additional muscle contractions.

Aim 3: To test the hypothesis that obesity induces an endothelial phenotype change that creates an environment for both EDD and exercise dysfunction. We propose that obesity alters endothelial enzymes which help explain the mechanistic changes in vasodilation.

Aim 4: To test the hypothesis that obesity elicits altered EDD and functional vasodilation due to altered functional potassium channel signaling. We propose that K+ channel function accounts for unexplained differences in EDD and functional vasodilation. More specifically, we hypothesize that inhibition of K+-mediated hyperpolarization (via inward rectifying K+ channels (KIR)) will identify differential vasodilator mechanisms between lean and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 - ≤ 40 years of age
* Blood pressure systolic ≤125 and diastolic ≤85 mmHg (Lean control) and <140 and diastolic <90 mmHg (Obese subjects)
* BMI <25 kg/m2 (Lean control) and ≥30 kg/m2 (Obese subjects)
* Fasting blood glucose <100 mg/dL
* Fasting LDL <130 mg/dL
* Fasting blood triglycerides <150 mg/dL
* Females: Premenopausal with a regular menstrual cycle. Negative pregnancy test. Note: Must be studied in the early follicular phase (day 1-5) of their menstrual cycle or the low hormone phase of oral contraceptive use.

Exclusion Criteria:

* Specific to obese subjects only (to exclude obese subjects with metabolic syndrome):

  a. If Systolic BP 130 ≤ BP < 140 mmHg or Diastolic BP 85 ≤ BP < 90 mmHg i. HDL < 40 mg/dL for men ii. HDL < 50 mg/dL for women
* Increased risk of bleeding
* Sensitivity to lidocaine
* Procoagulant or other clotting disorders
* Taking cardiovascular medications (anti-hypertensives, statins, platelet inhibitors, etc.) or metabolic medications (insulin-sensitizing)
* Regularly (≥5 days/week) take acetylsalicylic acid and/or non-steroidal anti-inflammatory drugs (NSAIDs)
* Self-reported current diagnosis of exhibiting obstructive sleep apnea
* Self-reported current or past diagnosis of diabetes
* Self-reported history of peripheral vascular disease
* Self-reported history of hepatic disease
* Self-reported history of renal disease
* Self-reported history of hematologic disease
* Self-reported history of stroke
* Current use of tobacco (i.e. smoke, smokeless, and vapor). Prior tobacco use with >1 year abstaining is allowed.
* Participation in vigorous aerobic exercise >90 minutes per week
* Arterial structures in the arm that are not conducive to study in the laboratory setting
* Females: Self-reported pregnancy and/or breastfeeding, diagnosed with polycystic ovarian syndrome, or without regular menses. Urine pregnancy test will be performed on study day to ensure subject is not pregnant on study day.
* An abnormality or contraindication to study participation which is not covered in the eligibility criteria.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04-16 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2021-11 (Actual)

PRIMARY OUTCOMES:
Change in limb blood flow in response to stimuli that cause vasodilation (ATP, ISO, BK, Ach, muscle contractions). | Through study completion
  Change in limb blood flow (ml/min), measured with Doppler ultrasound, in response potassium vasodilation (EDD or ROV). The change in blood flow will be calculated by taking the difference between the stimulus blood flow response and the baseline blood flow. These changes will be compared between lean and obese.
Change in limb blood flow in response to barium chloride infusion which inhibits potassium channel vasodilation. | Through study completion
  Change in limb blood flow (ml/min), measured with Doppler ultrasound, in response to barium chloride infusion (inhibition of K+ vasodilation). This will be calculated by taking the difference between the stimulus blood flow response and the stimulus blood flow response in the presence of barium chloride. These changes will be compared between lean and obese.

SECONDARY OUTCOMES:
Endothelial cell collection from arterial catheter to measure protein expression. | Through study completion
  Protein expression in endothelial cells harvested from arterial catheter that may be responsible for EDD or ROV functional changes (optional for subjects). Immunohistochemical methods will be used. Differences in protein expression will be assessed semi-quantitatively by normalizing expression to standard human endothelial cell cultures.
Change in blood flow in response to L-NMMA and ketorolac in the presence of barium chloride | Minutes/seconds between baseline and peak response to stimuli
  Change in limb blood flow (ml/min), measured with Doppler ultrasound, in response to L-NMMA and ketorolac infusion in the presence of barium chloride infusion. This will be calculated by taking the difference between the stimulus blood flow response and the stimulus blood flow response in the presence of all inhibitors (barium chloride, ketorolac, and L-NMAA). These changes will be compared between lean and obese.

CONTACTS AND LOCATIONS:
Overall Officials: William Schrage, Ph.D., Principal Investigator — UW Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No